CLINICAL TRIAL: NCT01369238
Title: Clinical Research on the Efficacy of East-West Collaborative Medicine Using Bee-Venom Acupuncture Therapy on Whiplash-Associated Disorders After Traffic Collisions; A Randomized, Controlled, Parallel Trial
Brief Title: East-West Collaborative Medicine Using Bee-Venom Acupuncture on Whiplash-Associated Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Pharmacoacupuncture Institute (Other)
Responsible Party: Chung, Su-Yeon/Academic Team, Korean Pharmacoacupuncture Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOMC 2010-04
Record Dates: First submitted 2011-05-12; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Whiplash Injuries
Keywords: bee venom acupuncture; east west collaborative medicine; whiplash associated disorder
MeSH Terms: conditions — Whiplash Injuries | interventions — Acupuncture Therapy; pyranoprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bee Venom Acupuncture & zaltoprofen (Experimental)
  Interventions: Device: Bee Venom Acupuncture Therapy; Drug: zaltoprofen
- zaltoprofen (Active Comparator)
  Interventions: Drug: zaltoprofen
- Bee Venom Acupuncture (Active Comparator)
  Interventions: Device: Bee Venom Acupuncture Therapy

INTERVENTIONS:
Device: Bee Venom Acupuncture Therapy — 1:4000, SC 1cc/day, 2~3days/wk, for 1 month
  Other Names: pharmacoacupuncture
  Arms: Bee Venom Acupuncture; Bee Venom Acupuncture & zaltoprofen
Drug: zaltoprofen — 80mg/Tab, per os 1Tab tid, for 2 months
  Other Names: soleton
  Arms: Bee Venom Acupuncture & zaltoprofen; zaltoprofen

SUMMARY:
1. Purpose of study

   1. To evaluate the efficacy of East-West collaborative medicine using Bee-Venom Acupuncture Therapy on Whiplash-Associated Disorders using VAS scale
   2. To evaluate the efficacy of East-West collaborative medicine using Bee-Venom Acupuncture Therapy on Whiplash-Associated Disorders using NDI, BDI, SF-36, and EQ-5D.
2. Interventions & Groups

   1. group 1: Bee-Venom Acupuncture Therapy
   2. group 2: zaltoprofen
   3. group 3: Bee-Venom Acupuncture Therapy & zaltoprofen

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Whiplash injuries
* Must have cervicalgia of more than VAS 5

Exclusion Criteria:

* cancer, osteoporosis, ankylosing spodylitis, cauda equina syndrome, infection
* spinal operation
* other musculoskeletal pain
* physicological or mental disorders

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
pain scores on Visual Analogue Scale | changes from baseline in VAS at 1 month

SECONDARY OUTCOMES:
neck disability scores on Neck Disability Index | changes from baseline in NDI at 1 month
depression scores on Beck Depression Inventory | changes from baseline in BDI at 1 month
quality of life scores on short form SF-36 | changes from baseline in short form SF-36 at 1 month
quality of life scores on EQ-5D | changes from baseline in EQ-5D at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Hee Chung, Study Chair — Kyung Hee Oriental Medical Center; Jun-Hwan Lee, Study Director — Kyung Hee University Hospital at Gangdong; Koh-Woon Kim, Principal Investigator — Kyung Hee Oriental Medical Center